CLINICAL TRIAL: NCT00068419
Title: A Phase II Study of Sulindac and Tamoxifen in Patients With Desmoid Tumors That Are Recurrent or Not Amenable to Standard Therapy
Brief Title: Sulindac and Tamoxifen in Treating Patients With Desmoid Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARST0321; NCI-2009-00424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000322260 (Other: PDQ (Physician Data Query)); COG-ARST0321 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2019-02

CONDITIONS: Desmoid Tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Tamoxifen; Sulindac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy, anti-estrogen therapy) (Experimental): Patients receive oral sulindac and oral tamoxifen citrate twice daily for up to 12 months (four 3-month courses) in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 1 additional month of treatment beyond documentation of CR.
  Interventions: Drug: tamoxifen citrate; Drug: sulindac; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tamoxifen citrate — Given orally
  Other Names: Nolvadex; TAM; tamoxifen; TMX
Drug: sulindac — Given orally
  Other Names: Aflodac; Algocetil; Clinoril; SULIN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving sulindac together with tamoxifen works in treating patients with desmoid tumor. Sulindac may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Hormone therapy using tamoxifen may fight cancer by blocking the use of estrogen. Combining sulindac with tamoxifen may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the safety and efficacy of sulindac and tamoxifen in patients with recurrent desmoid tumor (DT) and primary DT that is not readily amenable to surgery or radiation therapy.

SECONDARY OBJECTIVES:

I. Determine the tumor response rate in patients treated with this regimen.

II. Correlate changes in Magnetic Resonance Imaging (MRI) signal features of the tumor with clinical outcome in patients treated with this regimen.

III. Correlate pathological studies of cyclooxygenase-2 (COX-2) and estrogen/progesterone receptor expression in the tumor with clinical outcome in patients treated with this regimen.

IV. Collect information about clinical factors that make a tumor unresectable at diagnosis and resectable during the four courses of study treatment.

V. Determine whether short-term endocrine toxicity is associated with treatment with this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sulindac and oral tamoxifen twice daily for up to 12 months (four 3-month courses) in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 1 additional month of treatment beyond documentation of CR.

After completion of study treatment, patients are followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed desmoid tumor, meeting 1 of the following criteria:

  * Newly diagnosed disease

    * Not previously treated
    * Not amenable to complete surgical resection and/or radiotherapy

      * If surgical resection was attempted, there must be gross residual disease measurable by MRI
  * Radiographically documented recurrent or progressive disease

    * No prior chemotherapy or radiotherapy for the present recurrence

      * Tumors that progressed on prior chemotherapy are allowed provided patients have not received chemotherapy for this recurrence
* Measurable disease by gadolinium-enhanced MRI
* No other fibroblastic lesions or fibromatoses

  * Lipofibromatosis or desmoplastic fibroma of the bone allowed
* Performance status - Karnofsky Score 50-100% (patients over age 16)
* Performance status - Lansky Score 50-100% (patients age 16 and under)
* At least 8 weeks
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 10.0 g/dL (transfusion allowed)
* No hemophilia
* No von Willebrand disease
* No other clinically significant bleeding diathesis
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alanine aminotransferase (ALT) less than 2.5 times ULN
* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* No prior deep venous thrombosis
* Electrocardiogram (EKG) normal
* Chest x-ray normal
* No prior significant gastrointestinal hemorrhage
* No prior peptic ulcer disease
* Not pregnant or nursing
* Fertile patients must use effective nonhormonal contraception
* No evidence of active graft-versus-host disease
* No allergy to aspirin
* Recovered from prior immunotherapy
* At least 7 days since prior anticancer biologic agents
* At least 6 months since prior allogeneic stem cell transplantation
* More than 1 week since prior growth factors
* No concurrent immunomodulating agents
* No prior nonsteroidal anti-inflammatory drugs (NSAIDs) for desmoid tumor
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No concurrent anticancer chemotherapy
* No prior estrogen antagonists for desmoid tumor
* No concurrent hormonal contraceptives
* No concurrent steroids except for non tumor indications (e.g., asthma or severe allergic reactions)
* No concurrent NSAIDs for desmoid tumor

  * Occasional NSAIDs for musculoskeletal or other pain are allowed
* Recovered from prior radiotherapy
* No concurrent adjuvant radiotherapy
* No concurrent participation in another COG therapeutic study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2004-02; Primary Completion 2010-04-26 (Actual); Study Completion 2010-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Skapek, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Started | 70
Completed | 10 (Participant flow data reported here are for the period of protocol therapy.)
Not Completed | 60
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 24
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 14
Not completed — Ineligible | 11

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 51
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 63
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Failure Free at 2 Years Following Study Entry
Description: Kaplan Meier estimate of failure free survival at 2 years, where failure free survival is defined as the time to relapse, progression, second malignancy, and death whichever occurs first.
Time Frame: Up to 2 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 59
percentage of participants | 36 [23 to 48]

2. Primary Outcome: Percentage of Patients Experiencing a Grade 3 or Higher Adverse Event During Therapy.
Description: The percentage of patients experiencing a grade 3 or higher adverse event as assessed by the National Cancer Institute Common Toxicity Terminology for Adverse Events v3.0
Time Frame: Up to 12 months
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 59
Percentage of participants | 3.4 [0 to 8.0]

3. Secondary Outcome: Percentage of Patients With Tumor Response From Imaging
Description: Percentage of patients with a tumor response where tumor response is assessed according to Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: Baseline up to 5 years
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 59
Percentage of participants | 8.0 [1.1 to 14.9]

4. Secondary Outcome: Mean Change in Response Measured by MRI
Description: The mean change in response measured by MRI. Response is assessed by the lesion size which is derived from the sum of the longest of the three orthogonal diameters (from MRI) of each target lesion.
Time Frame: From baseline to up to 5 years
Population: Outcome not reported because the required data were not recorded.
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Patients Failure Free at 2 Years by Pathological Response
Description: The failure free survival is compared by the log-rank test between patient subgroups defined by pathological response of cyclooxygenase-2 (COX-2) and estrogen/progesterone receptor expression
Time Frame: From enrollment to up to 2 years
Population: Data not available for analysis due to no data were collected
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Patients Experiencing Short-term Endocrine Toxicity
Description: The percentage of patients experiencing short-term endocrine toxicity between treatment groups is compared using the chi-square test
Time Frame: At study entry
Population: Data not available for analysis due to no data were collected.
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of protocol therapy plus 30 days.
Description: Reporting is for all patients who received protocol therapy (11 patients were ineligible for protocol therapy).
Arm/Group | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy)
Serious Adverse Events (participants affected / at risk) | 2/59
Other Adverse Events (participants affected / at risk) | 42/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy) (N=59)
Abdominal pain (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy, Anti-estrogen Therapy) (N=59)
Abdominal pain (Gastrointestinal disorders) | 20
Acidosis (Metabolism and nutrition disorders) | 2
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 7
Ataxia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood gonadotrophin abnormal (Investigations) | 2
Catheter related infection (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 2
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 7
Endocrine disorders - Other (Endocrine disorders) | 3
Esophagitis (Gastrointestinal disorders) | 1
Eye disorders - Other (Eye disorders) | 5
Fatigue (General disorders) | 8
Fever (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Flushing (Vascular disorders) | 1
Gait disturbance (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
GGT increased (Investigations) | 1
Gynecomastia (Reproductive system and breast disorders) | 1
Headache (Nervous system disorders) | 12
Hearing impaired (Ear and labyrinth disorders) | 1
Hot flashes (Vascular disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Investigations - Other (Investigations) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 4
Non-cardiac chest pain (General disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 3
Serum amylase increased (Investigations) | 1
Sinusitis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Stomach pain (Gastrointestinal disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vascular disorders - Other (Vascular disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.